CLINICAL TRIAL: NCT06261346
Title: Safety and Efficacy of Brief Intraoperative Corneal Endothelial Graft Incubation in Plasma Rich in Growth Factors (PRGF) for Reducing Postoperative Endothelial Cell Loss
Brief Title: Plasma Rich in Growth Factors in Corneal Endothelial Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Florida lions eye bank (Unknown)
Responsible Party: Principal Investigator, Alfonso Sabater, Associate Professor of Clinical Ophthalmology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20230420
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Fuchs' Endothelial Dystrophy; Corneal Edema
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Edema | interventions — Descemet Stripping Endothelial Keratoplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRGF group (Experimental): Participants tissue will be incubated in plasma rich in growth factors prior to endothelial keratoplasty procedure. Participants will be followed up for up to 1 year.
  Interventions: Procedure: Endothelial keratoplasty; Biological: PRGF
- Control group (Active Comparator): Participants will undergo endothelial keratoplasty procedure. Participants will be followed up for up to 1 year.
  Interventions: Procedure: Endothelial keratoplasty

INTERVENTIONS:
Procedure: Endothelial keratoplasty — Surgical replacement of the corneal endothelial cell layer (the cell layer lining the inner surface of the cornea) with brief incubation of the donor tissue in PRGF prior to graft implantation. This incubation will be a one time procedure done to the tissue in the operating room.
  The endothelial keratoplasty is 30-45 minutes.
Biological: PRGF — Plasma Rich in Growth Factors (PRGF) is a mixture of proteins and growth factors obtained from the blood of the patient.
  PRGF incubation lasts 15 minutes. It is a one-time procedure performed on the tissue that will be done in the operating room prior to endothelial keratoplasty.
  Arms: PRGF group

SUMMARY:
The purpose of the study is to determine the safety and efficacy of brief intraoperative corneal endothelial graft incubation in plasma rich in growth factors (PRGF) for reducing postoperative endothelial cell loss.

ELIGIBILITY:
Inclusion Criteria:

* undergoing endothelial keratoplasty (DSEK or DMEK) at the Bascom Palmer Eye Institute or Price Vision Group, using corneal graft tissue within 14 days of preservation

Exclusion Criteria:

* History of corneal transplantation in the study eye, Best corrected visual acuity (BCVA) worse than 20/40 in the contralateral eye, systemic immunosuppression, previous intraocular surgical procedures (other than cataract surgery) such as glaucoma tubes or silicone oil.

The following special populations will be excluded.

* Adults unable to consent
* Pregnant women
* Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in endothelial cell percentage | Baseline, 6 months
  Central corneal endothelial cell percentage will be assessed by specular microscopy and compared with the baseline donor endothelial cell percentage measured by the provider eye bank to determine endothelial cell changes.

SECONDARY OUTCOMES:
Corneal endothelial cell density | Up to 12 months
  Central corneal endothelial cell density by specular microscopy (cells/millimeter^2)
Change in Endothelial cell density | Baseline, up to 12 months
  Change in central corneal endothelial cell density will be assessed by specular microscopy (cells/millimeter^2) and compared with the baseline donor endothelial cell density reported by the provider eye bank to determine endothelial cell loss
Visual acuity measured by snellen chart | Up to 12 months
  Participants will have their best corrected visual acuity measured as values expressed using the Snellen chart.
Number of re-bubbling for graft attachment | Up to 2 months
  The number of air re-injections for graft attachment within the first 2 months will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso L Sabater, MD, Principal Investigator — Bascom Palmer Eye Institute
Locations (2):
- United States (2):
  - Bascom Palmer Eye Institute, Miami, Florida
  - Price Vision Group, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No